CLINICAL TRIAL: NCT00695422
Title: A Companion Protocol to Evaluate Anogenital Human Papillomavirus (HPV) Infection and Anogenital Squamous Intraepithelial Lesions (ASIL) in Subjects Participating in AMC Clinical Trials
Brief Title: Detecting Anal and Genital Human Papillomavirus Infection and Squamous Intraepithelial Lesions in HIV-Positive Patients Enrolled in AIDS Cancer Clinical Trials
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AMC-058; U01CA121947 (NIH); CDR0000590397 (Other: NCI)
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Aids-related Malignancies; Lymphoma; Precancerous Condition; Sarcoma
Keywords: high-grade squamous intraepithelial lesion; low-grade squamous intraepithelial lesion; human papilloma virus infection; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related Kaposi sarcoma; AIDS-related lymphoblastic lymphoma; AIDS-related malignancies; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; multicentric Castleman disease; HIV Infections
MeSH Terms: conditions — Lymphoma; Precancerous Conditions; Sarcoma; Squamous Intraepithelial Lesions; Papillomavirus Infections; AIDS-related Kaposi sarcoma; Multi-centric Castleman's Disease; HIV Infections | interventions — Polymerase Chain Reaction; Histological Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens, anal cytology and biopsy of any lesions observed, cervical cytology and biopsy of any lesions observed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Specimen Collection: Blood collection, anal cytology and biopsy of observed lesions. Additional cervical cytology and biopsy for females.
  Interventions: Genetic: polymerase chain reaction; Other: cytology specimen collection procedure; Other: histological technique; Procedure: colposcopic biopsy

INTERVENTIONS:
Genetic: polymerase chain reaction — PCR for HPV DNA detection, performed on specimens collected at baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol.
Other: cytology specimen collection procedure — Detection of HPV-associated neoplasia at baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol.
Other: histological technique — Detection of HPV-associated neoplasia at baseline, treatment discontinuation on parent protocol, final visit on parent protocol.
Procedure: colposcopic biopsy — Where observed during HRA, collection of tissue for detection of HPV-associated neoplasia at baseline, treatment discontinuation on parent protocol, final visit on parent protocol.

SUMMARY:
RATIONALE: Diagnostic procedures, such as anal swab collection, digital rectal examination, and anal endoscopy and biopsy, may help find and diagnose anal and genital human papillomavirus infection and squamous intraepithelial lesions and help doctors plan better treatment.

PURPOSE: This clinical trial is studying ways to detect anal and genital human papillomavirus infection and squamous intraepithelial lesions in HIV-positive patients enrolled in an AIDS cancer clinical trial.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if various pharmacotherapeutic agents investigated in primary AIDS Malignancy Clinical Trials (AMC) for diseases other than human papillomavirus (HPV)-associated neoplasia have any preliminary evidence of activity against anogenital HPV infection or anogenital squamous intraepithelial lesions (ASIL) in HIV-positive patients participating in these trials.
* To describe changes in the types of anal HPV present and the prevalence of ASIL in patients treated on these studies.
* To evaluate cervical HPV infection and cervical/vulvovaginal disease in HIV-positive women participating in these trials.
* To describe changes in cervical HPV infection and cervical/vulvovaginal disease in these women after undergoing various study treatments.

OUTLINE: This is a multicenter study.

Patients undergo anal swab collection at baseline to obtain samples for anal cytology, anal human papillomavirus (HPV) typing, and other HPV-related testing (e.g., HPV viral load). Digital rectal examinations (DRE) are also performed as part of the baseline physical examination. Female patients also undergo cervical swab collection for cervical HPV testing and cytology, as well as colposcopy (if available) of the cervix and vulvovaginal region to completely assess lower genital tract HPV-related lesions. At sites where high-resolution anoscopy (HRA) is available, patients are encouraged, but not required, to have an HRA with biopsy of any visualized lesions within 30 days of collection of the swabs.

After baseline assessments, patients undergo treatment with the investigative agent according to the study protocol requirements. If study treatment continues beyond 6 months, additional anal and cervical swabs are obtained for anal and cervical HPV and cytology along with DREs every 6 months until completion of study treatment and at the final study visit. Patients may also undergo additional HRA with biopsy and/or colposcopy of the lower genital tract with biopsy (women only) at this time. Patients with an abnormal anal cytology or histology are referred for HRA per local standard of care. If HRA is not available at the treatment site, patients undergo a DRE, and those with an abnormal DRE are referred for evaluation by a surgeon.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Serologic documentation of HIV infection by any FDA-approved tests
* Enrolled in an AIDS Malignancy Clinical Trials Consortium (AMC) clinical trial of any new or existing pharmacotherapeutic agent for treatment of disease other than human papillomavirus (HPV)-associated neoplasia

  * AMC study must have an accrual target of > 15 patients

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 60-100%
* Life expectancy ≥ 3 months
* Not pregnant or nursing
* Patients receiving myelosuppressive therapy must meet the following criteria:

  * ANC > 1,000/μL
  * Platelet count > 50,000/μL
  * Evaluated before treatment or completely recovered from their nadir
* Able to understand and willing to sign a written informed consent document
* No bleeding disorder or requirement for anticoagulation that would contraindicate any biopsy of the anal canal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients who are study participants on interventional AMC protocols for diseases other than HPV-associated neoplasia with an accrual goal of 15 patients or more.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2008-05-14 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Activity of pharmacotherapeutic agents being investigated in AIDS Malignancy Clinical Trials (AMC) against anogenital human papillomavirus (HPV) infection or anogenital squamous intraepithelial lesions (ASIL) | Baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol
Cervical HPV infection and cervical/vulvovaginal disease in women participating in AMC clinical trials | Baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol
Changes in cervical HPV infection and cervical/vulvovaginal disease after treatment on AMC studies | Baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol
Changes in anal HPV types present | Baseline, every 6 months while on parent protocol, treatment discontinuation on parent protocol, final visit on parent protocol
Frequency of ASIL | Baseline, treatment discontinuation on parent protocol, final visit on parent protocol

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Berry, MD, Principal Investigator — University of California, San Francisco
Locations (10):
- United States (10):
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Baylor University Medical Center - Houston, Houston, Texas
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No